CLINICAL TRIAL: NCT01964014
Title: Clinical Investigation for Safety and Efficacy, Patient Reported Outcomes of the Conversion to ONce-a-day Immunosuppression After Kidney Transplantation
Brief Title: Once-a-day Immunosuppression(CISECON_a_day)
Acronym: CISECON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Chang kwon oh, Professor,Department of surgery, Ajou University School of Medicine, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-CT4-11-391
Record Dates: First submitted 2013-10-01; First posted 2013-10-17 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Renal Disease
Keywords: once
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- advagraf (Experimental): The same capacity advagaf + sirolimus
  Interventions: Drug: advagrf

INTERVENTIONS:
Drug: advagrf — All enrolled subjects will discontinue the existing Tacrolimus preparations for 6 months from enrollment and be converted to Extended Release Tacrolimus at a biologically equivalent dose. They will also discontinue enteric-coated mycophenolate sdium or mycophenolate sodium and be treated with Sirolimus and observed.
  advagrf+sirolimus one time to eat.

SUMMARY:
The objective of this study is to assess the efficacy and safety and Immunosuppressant Therapy Barrier Scale (ITBS) of once daily immunosuppressant maintenance therapy in patients who had kidney transplantations earlier.

DETAILED DESCRIPTION:
This is a 6-month, single-arm, multi-center, open-label, continuous cohort study. 160 subjects who had kidney transplantations at least 3 months earlier will participate in the study. All enrolled subjects will discontinue the existing Tacrolimus preparations for 6 months from enrollment and be converted to Extended Release Tacrolimus at a biologically equivalent dose. They will also discontinue enteric-coated mycophenolate sdium or mycophenolate sodium and be treated with Sirolimus and observed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at the age of 20 to 65 who had kidney transplantations at least 3 months ago.
* Recipients of kidney transplantations from a deceased / cadaveric donor, non-heart beating cadaveric donor / organ donor after cardiac death, or non-blood related or blood related live donor.
* Patients being treated with Tacrolimus or Extended Release Tacrolimus as the existing immunosuppressant maintenance therapy.
* Able and willing to give informed consent to study participation, having signed the informed consent form according to appropriate procedures, and capable of participating in the study by making visits according to study plans.

Exclusion Criteria:

* HIV, HBsAg, or anti-HCV test positive patients or having received kidney transplantations from an HIV, HBsAg, or anti-HCV test positive donor.
* History of severe allergies or hypersensitivities to drugs used in the study or other drugs with a similar chemical structure requiring acute (within the past 4 weeks) or chronic treatment.
* Having received other investigational product within 30 days prior to enrollment into this study.
* Women of childbearing potential who plan to become pregnant, pregnant and/or lactating women, women who do not intend to use effective contraceptives.
* Having uncontrolled diseases or medical conditions requiring continuous treatment.
* History of alcohol or drug addiction within the past 3 months or incapable of appropriate communications due to reasons such as mental illness.
* Absolute neutrophil count <1,500/mm3 or leukocyte count <2,500/mm3 or platelet count <75,000/mm3 at screening or severe metabolic disorders (including functional disorders).
* Having experienced the following condition within the past 1 month:

  * Serum creatinine > 2.0 mg/dl more than twice.
  * 24 hr urine protein≥750 mg/day
  * Diagnosed with or treated for a rejection reaction or an infection or hospitalized due to other medical reasons.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
acute rejection reaction treated or confirmed by biopsy, loss of graft, death, or lost to follow-up | 6months
  The primary objective of this study is to investigate the efficacy of Advagraf ® (Extended Release Tacrolimus) at 6 months after immunosuppressant conversion to the once daily therapy. The efficacy is defined as the incidence rate of composite endpoints of efficacy failure (acute rejection reaction treated or confirmed by biopsy, loss of graft, death, or lost to follow-up).

SECONDARY OUTCOMES:
renal functions | 6months
  Difference in renal functions (eGFR by MDRD method), urine protein excretion and P/C ratio (A/C ratio), transplant kidney biopsy histology (if biopsy is performed).
serious adverse events | 6months
  Frequency and severity of adverse events and serious adverse events
cardiovascular health | 6months
  Treatment impact on cardiovascular health: blood pressure and cardiovascular events (acute myocardial infarction, unstable angina pectoris, heart failure, stroke).
NODAT | 6months
  Incidence rate of new onset diabetes after transplantation (NODAT) requiring treatment.
hematology issue | 6months
  Frequency of anemia, leucopenia, and thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: chang-kwon oh, M.D.,Ph.D., Principal Investigator — Ajou University School of Medicine
Locations (7):
- South Korea (7):
  - Nephrology, Pusan National University Hospital, Busan
  - Bundang CHA Medical Center,, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Gyeonggido
  - Korea University Medical Center, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hosptial, Seoul
  - Dept. of Surgery, Ulsan University Hospital, Ulsan